CLINICAL TRIAL: NCT07175571
Title: Prospective Randomized Sibling-Oocyte Trial Comparing Fertilization and Embryo Development Outcomes Between Intracytoplasmic Sperm Injection (ICSI) and Conventional IVF Using Frozen Donor Sperm
Brief Title: SISTER: Sibling Oocyte Insemination With Frozen Sperm From Third Party Donors: Evaluation of Reproductive Techniques
Acronym: SISTER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shady Grove Fertility Reproductive Science Center (Other)
Responsible Party: Principal Investigator, Kate Devine, Medical Director and Chief Research Officer, Shady Grove Fertility Reproductive Science Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SISTER Study
Record Dates: First submitted 2025-09-09; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-05

CONDITIONS: Infertility, Female; Reproductive Techniques, Assisted; Fertilization in Vitro
Keywords: Intracytoplasmic Sperm Injection (ICSI); Conventional IVF; Frozen Donor Sperm; Sibling-Oocyte Design; Non-Male Factor Infertility; Blastulation Rate; Total Fertilization Failure (TFF); Fertilization Outcomes; Embryo Quality; Clinical Pregnancy Rate; Assisted Reproductive Technology (ART); Embryo Development; In Vitro Fertilization; Oocyte Randomization; Female Infertility; Cryopreserved Sperm; Randomized Controlled Trial (RCT); Reproductive Medicine; Fertility Treatment
MeSH Terms: conditions — Infertility, Female; Helping Behavior | interventions — Sperm Injections, Intracytoplasmic

STUDY DESIGN:
Intervention Model Description: This is a randomized sibling-oocyte controlled trial in which each participant's retrieved oocytes are split between two insemination methods: intracytoplasmic sperm injection (ICSI) and conventional in vitro fertilization (IVF). Randomization occurs at the oocyte level, not at the participant level. For participants with an even number of mature oocytes, half are randomly assigned to ICSI and half to conventional IVF. For participants with an odd number, the extra oocyte is randomly allocated using a pre-specified scheme. This within-subject design allows direct comparison of fertilization and embryo development outcomes between the two methods while minimizing inter-patient variability.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intracytoplasmic Sperm Injection (ICSI) (Experimental): In this arm, a portion of each participant's mature oocytes will be inseminated using intracytoplasmic sperm injection (ICSI). A single frozen-thawed donor sperm cell will be injected directly into each oocyte using micromanipulation techniques. The oocyte assignment to ICSI will be determined through randomized sibling-oocyte allocation. Embryos will be cultured under standard laboratory conditions and assessed for fertilization (2PN), blastulation, embryo quality, and early clinical pregnancy outcomes.
  Interventions: Procedure: Intracytoplasmic Sperm Injection (ICSI)
- Conventional Insemination (IVF) (Experimental): In this arm, a portion of each participant's oocytes will be inseminated using the conventional in vitro fertilization (IVF) method. Frozen-thawed donor sperm with normal post-thaw parameters will be co-incubated with oocytes in culture media for fertilization. The oocyte assignment to this method will be determined through randomized sibling-oocyte allocation. Embryos will be cultured under the same laboratory conditions and assessed for fertilization (2PN), blastulation, embryo quality, and early clinical pregnancy outcomes.
  Interventions: Procedure: Conventional Insemination (IVF)

INTERVENTIONS:
Procedure: Intracytoplasmic Sperm Injection (ICSI) — Mature oocytes are injected with a single frozen-thawed donor sperm cell using micromanipulation under a microscope. This fertilization method is performed shortly after oocyte retrieval. Sperm used are pre-screened and standardized for post-thaw motility and morphology. ICSI is conducted in accordance with standard embryology lab protocols. The oocyte allocation to ICSI is randomized within each participant's cycle.
  Arms: Intracytoplasmic Sperm Injection (ICSI)
Procedure: Conventional Insemination (IVF) — Oocytes are inseminated by co-incubation with frozen-thawed donor sperm in a culture dish for 16-18 hours. Sperm are washed and prepared according to lab protocol to ensure motility and concentration suitability. This method does not involve direct sperm injection. Oocytes are randomly assigned to this method within each participant's retrieved cohort.
  Arms: Conventional Insemination (IVF)

SUMMARY:
The goal of this clinical trial is to learn whether two different methods of helping eggs and sperm join-intracytoplasmic sperm injection (ICSI) and conventional in vitro fertilization (IVF)-lead to better embryo development when using frozen donor sperm in people who do not have male fertility problems. The main questions it aims to answer are:

Does one method create more usable embryos (blastocysts) than the other?

Is there a difference in how often fertilization does not happen at all?

Do either of the methods lead to better embryo quality or early pregnancy?

Participants will:

Have their eggs divided into two groups. One group will be fertilized using ICSI (where a sperm is injected directly into an egg), and the other using conventional IVF (where eggs are mixed with sperm in a dish).

The fertilization method for each egg will be randomly assigned, with a random process also used to determine the assignment of any extra egg when an odd number is collected.

Continue regular fertility treatment while the study team compares the results of each fertilization method.

This study includes people with non-male factor infertility and uses frozen donor sperm. It hopes to learn whether ICSI, which is often used even when it may not be needed, truly helps improve outcomes compared to conventional IVF in these cases.

DETAILED DESCRIPTION:
This is a prospective, randomized sibling-oocyte controlled trial designed to compare fertilization and embryo development outcomes between intracytoplasmic sperm injection (ICSI) and conventional in vitro fertilization (IVF) using cryopreserved donor sperm in non-male factor infertility cycles. Despite widespread use of ICSI in assisted reproductive technology (ART), there is insufficient evidence supporting its routine use in non-male factor indications, especially in cycles utilizing frozen sperm where male factor infertility is not a contributing variable.

The study aims to address ongoing clinical debate and practice variation by evaluating whether ICSI offers meaningful advantages over conventional IVF in this specific context. Previous retrospective and meta-analytic data have suggested that while ICSI may reduce total fertilization failure (TFF), it may not improve-and may even negatively impact-other key clinical outcomes such as blastulation rate, embryo quality, and early pregnancy rates in non-male factor populations. Additionally, concerns about increased pregnancy-related complications with ICSI have been raised.

To reduce inter-patient variability and enhance internal validity, a sibling-oocyte design will be employed, allowing within-patient comparison of insemination methods. Oocytes retrieved from each participant will be randomized to either ICSI or conventional IVF. Randomization will be conducted prior to oocyte retrieval using computer-generated allocation. For patients with an even number of mature oocytes, half will be assigned to each insemination method. For those with an odd number, the extra oocyte will be randomly allocated according to the pre-specified scheme.

The fertilization process will begin shortly after oocyte retrieval. In the conventional IVF arm, mature oocytes will be inseminated using washed frozen-thawed donor sperm at a standard concentration and co-incubated for 16-18 hours. In the ICSI arm, a single motile sperm will be injected directly into each mature oocyte. All oocytes will undergo standard embryological assessment post-insemination, and embryos will be cultured under identical conditions.

The primary endpoint is the blastulation rate, defined as the number of usable blastocysts (meeting lab criteria for cryopreservation or transfer) per number of oocytes inseminated in each arm. Secondary outcomes include:

* Fertilization rate: number of 2PN zygotes per oocyte inseminated
* Incidence of TFF: no oocytes fertilized in a given arm
* Proportion of high-quality blastocysts, defined as grade BB or higher
* Early clinical pregnancy rate, as determined by ultrasound-confirmed intrauterine gestation Statistical analysis will use generalized estimating equations (GEE) for the primary outcome at the oocyte level to account for clustering within patients. Secondary outcomes will be analyzed using chi-square or Fisher's exact tests as appropriate. All data will be analyzed on an intention-to-treat basis.

The study will enroll approximately 178 participants over 12 months at Shady Grove Fertility, where frozen donor sperm with normal post-thaw parameters is routinely available. Only non-male factor infertility patients using frozen donor sperm will be eligible, ensuring a controlled sperm quality baseline across study arms.

The hypothesis is that conventional IVF will demonstrate equivalent or superior blastulation rates compared to ICSI, with non-inferior fertilization outcomes and potentially better embryo morphology. Results from this trial will help refine clinical guidelines and may support a more evidence-based, resource-efficient use of ICSI.

IRB approval has been obtained, and informed consent will be secured from all participants. All procedures will adhere to Good Clinical Practice and applicable regulatory guidelines. Data confidentiality will be maintained throughout.

ELIGIBILITY:
Inclusion Criteria:

* Female patients undergoing IVF with frozen donor sperm at Shady Grove Fertility Center
* Normal ovarian reserve (AMH > 1 ng/mL, AFC > 10)
* Absence of male factor infertility
* Post-wash parameters: >50% motility, >5mil concentration
* > 4 oocytes retrieved at time of transvaginal oocyte retrieval

Exclusion Criteria:

* Donor Sperm with significant male factor infertility (e.g., abnormal sperm concentration, motility, or morphology)
* Any medical condition contraindicating ART

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 95 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Blastulation Rate | Day 5 to Day 7 post-insemination
  The blastulation rate is defined as the number of "usable" blastocysts divided by the number of oocytes inseminated in each arm (ICSI and conventional IVF). A blastocyst is considered "usable" if it meets laboratory criteria for either cryopreservation or embryo transfer. Assessment is performed on Days 5-7 after fertilization using standard morphological grading under light microscopy.

SECONDARY OUTCOMES:
Fertilization Rate | Approximately 16-18 hours post-insemination
  The fertilization rate is the number of oocytes that develop two pronuclei (2PN), indicating successful fertilization, divided by the total number of oocytes inseminated. Oocytes are assessed approximately 16-18 hours after insemination. A 2PN zygote is a marker of normal fertilization in IVF/ICSI cycles.
Total Fertilization Failure (TFF) | Approximately 16-18 hours post-insemination
  TFF is defined as the percentage of insemination arms (either ICSI or conventional IVF) within a cycle that result in zero fertilized oocytes (0% 2PN). This is assessed at the patient level. For example, if none of the oocytes in the conventional IVF group fertilize, that arm is considered to have experienced TFF.
Proportion of High-Quality Blastocysts | Day 5 to Day 7 post-insemination
  This outcome measures the proportion of blastocysts graded BB or higher on standard morphological grading scales. Embryos are assessed on Days 5-7 post-insemination. Blastocyst quality is determined based on expansion, inner cell mass, and trophectoderm appearance. Only embryos reaching the blastocyst stage are included in this metric.
Early Clinical Pregnancy Rate | Approximately 5 to 7 weeks after embryo transfer
  Early clinical pregnancy is confirmed by the presence of a gestational sac visualized on transvaginal ultrasound, typically around 5-7 weeks after embryo transfer. The rate is calculated as the percentage of embryo transfer cycles in which at least one intrauterine pregnancy is confirmed.

CONTACTS AND LOCATIONS:
Overall Officials: Kate Devine, MD, Study Chair — Shady Grove Fertility
Locations (1):
- Shady Grove Fertility Rockville, Rockville, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Romero-Galisteo RP, Pinero-Pinto E, Palomo-Carrion R, Luque-Moreno C, Molina-Torres G, Gonzalez-Sanchez M. Translation, cross-cultural adaptation and validation of the Rett syndrome motor evaluation scale (RESMES): Spanish version. Eur J Paediatr Neurol. 2023 Nov;47:72-79. doi: 10.1016/j.ejpn.2023.09.008. Epub 2023 Sep 28. PMID 37788534
- [Background] Palermo G, Joris H, Devroey P, Van Steirteghem AC. Pregnancies after intracytoplasmic injection of single spermatozoon into an oocyte. Lancet. 1992 Jul 4;340(8810):17-8. doi: 10.1016/0140-6736(92)92425-f. PMID 1351601
- [Background] Hao G, Zhou X, Yan H, Wang X, Qiao L, Ni D, Shu W, Yu T. Emotional experience elicited by direct electrical stimulation: Case series and literature review. Epilepsia Open. 2023 Jun;8(2):547-558. doi: 10.1002/epi4.12729. Epub 2023 Apr 4. PMID 36932033
- [Background] Mao Z, Yao H, Zou Q, Zhang W, Dong Y. Digital Contact Tracing Based on a Graph Database Algorithm for Emergency Management During the COVID-19 Epidemic: Case Study. JMIR Mhealth Uhealth. 2021 Jan 22;9(1):e26836. doi: 10.2196/26836. PMID 33460389
- [Background] Teodorescu M, Barnet JH, Hagen EW, Palta M, Young TB, Peppard PE. Association between asthma and risk of developing obstructive sleep apnea. JAMA. 2015 Jan 13;313(2):156-64. doi: 10.1001/jama.2014.17822. PMID 25585327
- [Background] Mo DY, Tang YM, Wu EY, Tang V. Theoretical model of investigating determinants for a successful Electronic Assessment System (EAS) in higher education. Educ Inf Technol (Dordr). 2022;27(9):12543-12566. doi: 10.1007/s10639-022-11098-1. Epub 2022 Jun 3. PMID 35676938
- [Background] Zhang R, Xu S, Yuan M, Guo L, Xie L, Liao Y, Xu Y, Fu X. An ultrasmall PVP-Fe-Cu-Ni-S nano-agent for synergistic cancer therapy through triggering ferroptosis and autophagy. Nanoscale. 2023 Aug 3;15(30):12598-12611. doi: 10.1039/d3nr02708b. PMID 37462439